CLINICAL TRIAL: NCT01966458
Title: A Prospective, Randomized, Controlled, Unblinded, Multi-Center Clinical Trial to Evaluate the HeartWare™ Ventricular Assist Device System for Destination Therapy of Advanced Heart Failure
Brief Title: A Clinical Trial to Evaluate the HeartWare™ Ventricular Assist System (ENDURANCE SUPPLEMENTAL TRIAL)
Acronym: DT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HW004-A
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HeartWare® VAS (HVAD) (Experimental): Implant of HeartWare® Ventricular Assist System
  Interventions: Device: HeartWare® VAS (HVAD)
- Control LVAD (Active Comparator): Implant of FDA-approved LVAD approved for destination therapy
  Interventions: Device: Control LVAD

INTERVENTIONS:
Device: HeartWare® VAS (HVAD) — The HeartWare® VAS is an implantable centrifugal pump that was designed to provide flows up to 10 L/min in a small device that is both lightweight and simple to use.
  Arms: HeartWare® VAS (HVAD)
Device: Control LVAD — Any FDA-approved LVAD for destination therapy.
  Arms: Control LVAD

SUMMARY:
This is a prospective, randomized, controlled, unblinded, multi-center evaluation of safety and efficacy in patients implanted with a HeartWare® HVAD who receive improved blood pressure management. Subjects have chronic Stage D or NYHA Class IIIB/IV left ventricular failure who have received and failed optimal medical therapy, and who are ineligible for cardiac transplantation.

DETAILED DESCRIPTION:
The study will evaluate non-inferiority of neurologic injury incidence in a new cohort of subjects receiving improved blood pressure management to a control group (i.e., any FDA-approved LVAD for destination therapy). Secondary endpoints include: a comparison of stroke/TIA incidence to a reference observed in the original IDE clinical trial (HW004) that did not specify improved blood pressure management; and non-inferiority of stroke-free success on the originally implanted device to the control group. Subjects will be randomized to HeartWare® HVAD or control LVAD in a 2:1 ratio. Each subject receiving the HeartWare® HVAD or control LVAD is followed to the primary and secondary endpoints at 12 months, with a subsequent follow-up period extending to 60 months post-implant.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥18 years of age at consent
2. Body Surface Area (BSA) ≥ 1.2 m2
3. Patients with advanced heart failure symptoms (Class IIIB or IV) who are: (patient must meet one of the following)a. On optimal medical management, including dietary salt restriction and diuretics, for at least 45 out of the last 60 days and are failing to respond; or b. In Class III or Class IV heart failure for at least 14 days, and dependent on intra-aortic balloon pump (IABP) for 7 days and/or inotropes for at least 14 days
4. Left ventricular ejection fraction ≤ 25%
5. LVAD implant is intended as destination therapy
6. Must be able to receive either the HeartWare® HVAD or control LVAD
7. Patient must agree to participate in and comply with an improved blood pressure management program, including maintenance of a patient diary.
8. Female patients of childbearing potential must agree to use adequate contraceptive precautions (defined as oral contraceptives, intrauterine devices, surgical contraceptives or a combination of condom and spermicide) for the duration of the study.
9. The patient or legally authorized representative has signed the informed consent form

Exclusion Criteria:

1. Body Mass Index (BMI) > 40
2. Existence of any ongoing mechanical circulatory support (MCS) other than an intra-aortic balloon pump (IABP)
3. Prior cardiac transplant.
4. History of confirmed, untreated abdominal or thoracic aortic aneurysm > 5 cm.
5. Cardiothoracic surgery within 30 days of randomization.
6. Acute myocardial infarction within 14 days of implant as diagnosed by ST or T wave changes on the ECG, diagnostic biomarkers, ongoing pain and hemodynamic abnormalities as described (Figure 2) in the guidelines published in ACC/AHA 2007 Guidelines for the Management of Patients with Unstable Angina/Non-ST-Elevation Myocardial Infarction ;.
7. Patients eligible for cardiac transplantation
8. On ventilator support for > 72 hours within the four days immediately prior to randomization and implant.
9. Pulmonary embolus within three weeks of randomization as documented by computed tomography (CT) scan or nuclear scan.
10. Symptomatic cerebrovascular disease, stroke within 180 days of randomization or > 80% stenosis of carotid or cranial vessels.
11. Uncorrected moderate to severe aortic insufficiency. Correction may include repair or bioprosthesis at the time of implant.
12. Severe right ventricular failure as defined by the anticipated need for right ventricular assist device (RVAD) support or extracorporeal membrane oxygenation (ECMO) at the time of screening/randomization or right atrial pressure > 20 mmHg on multiple inotropes or right ventricular ejection fraction (RVEF) <15% with clinical signs of severe right heart failure (e.g. Lower extremity edema, ascites or pleural effusions refractory to treatment with diuretics and two inotropic drugs).
13. Active, uncontrolled infection diagnosed by a combination of clinical symptoms and laboratory testing, including but not limited to, continued positive cultures, elevated temperature and white blood cell (WBC) count, hypotension, tachycardia, generalized malaise despite appropriate antibiotic, antiviral or antifungal treatment.
14. Uncorrected thrombocytopenia or generalized coagulopathy (e.g., platelet count < 75,000, INR > 2.0 or PTT > 2.5 times control in the absence of anticoagulation therapy).
15. Intolerance to anticoagulant or antiplatelet therapies or any other peri- or postoperative therapy that the investigator may administer based upon the patient's health status.
16. Serum creatinine > 3.0 mg/dL within 72 hours of randomization or requiring dialysis or ultrafiltration.
17. Specific liver enzymes [AST (SGOT) and ALT (SGPT] > 3 times upper limit of normal within 72 hours of randomization.
18. A total bilirubin > 3 mg/dl within 72 hours of randomization, or biopsy proven liver cirrhosis or portal hypertension.
19. Pulmonary vascular resistance is demonstrated to be unresponsive to pharmacological manipulation and the PVR > 6 Wood units.
20. Patients with a mechanical heart valve.
21. Etiology of heart failure is due to, or associated with, uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis, active myocarditis or restrictive cardiomyopathy
22. History of severe COPD or severe restrictive lung disease (e.g. FEV1 <50%)
23. Participation in any other study involving investigational drugs or devices
24. Severe illness, other than heart disease, which would limit survival to < 3 years
25. Peripheral vascular disease with rest pain or ischemic ulcers of the extremities
26. Pregnancy
27. Patient unwilling or unable to comply with study requirements
28. Technical obstacles, which pose an inordinately high surgical risk, in the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Pagani, MD, Principal Investigator — University of Michigan Hospital; Joseph Rogers, MD, Principal Investigator — Duke University
Locations (47):
- United States (47):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic (Arizona), Phoenix, Arizona
  - The University of Southern California, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida Gainesville, Gainesville, Florida
  - University of Miami / Jackson Memorial Hospital, Miami, Florida
  - Tampa Transplant Institute/Tampa General Hospital, Tampa, Florida
  - The Emory Clinic Inc., Atlanta, Georgia
  - Saint Joseph Hospital of Atlanta, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - IU Health Methodist, Indianapolis, Indiana
  - St. Vincent Health, Indianapolis, Indiana
  - Jewish Hospital, Louisville, Kentucky
  - John Ochsner Heart & Vascular Institute, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Abbott Northwestern, Minneapolis, Minnesota
  - Mayo Clinic / St. Marys Hospital, Rochester, Minnesota
  - Washington University / Barnes Jewish Hospital, St Louis, Missouri
  - New York Presbyterian Hospital/Columbia, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundatiojn, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Heart Institute, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Northwest Cardiothoracic &Transplant Surgeons, Spokane, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Mahr C, McGee E Jr, Cheung A, Mokadam NA, Strueber M, Slaughter MS, Danter MR, Levy WC, Cheng RK, Beckman JA, May DM, Ismyrloglou E, Tsintzos SI, Silvestry SC. Cost-Effectiveness of Thoracotomy Approach for the Implantation of a Centrifugal Left Ventricular Assist Device. ASAIO J. 2020 Aug;66(8):855-861. doi: 10.1097/MAT.0000000000001209. PMID 32740343
- [Derived] Silvestry SC, Mahr C, Slaughter MS, Levy WC, Cheng RK, May DM, Ismyrloglou E, Tsintzos SI, Tuttle E, Cook K, Birk E, Gomes A, Graham S, Cotts WG. Cost-Effectiveness of a Small Intrapericardial Centrifugal Left Ventricular Assist Device. ASAIO J. 2020 Aug;66(8):862-870. doi: 10.1097/MAT.0000000000001211. PMID 32740129
- [Derived] Milano CA, Rogers JG, Tatooles AJ, Bhat G, Slaughter MS, Birks EJ, Mokadam NA, Mahr C, Miller JS, Markham DW, Jeevanandam V, Uriel N, Aaronson KD, Vassiliades TA, Pagani FD; ENDURANCE Investigators. HVAD: The ENDURANCE Supplemental Trial. JACC Heart Fail. 2018 Sep;6(9):792-802. doi: 10.1016/j.jchf.2018.05.012. Epub 2018 Jul 11. PMID 30007559

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were considered enrolled upon signing informed consent. 19 enrolled subjects weren't randomized as they were considered screen failures. 10 subjects were randomized but didn't receive a device due to death (with 1 subject dying post anesthesia but prior to Left Ventricular Assist Device (LVAD) implant) or screen failure prior to implant.
Groups:
- HeartWare® Ventricular Assist System (VAS): HeartWare® Ventricular Assist System (VAS): The HeartWare® VAS is an implantable centrifugal pump that was designed to provide flows up to 10 L/min in a small device that is both lightweight and simple to use.
- Control Left Ventricular Assist Device (LVAD): Control Left Ventricular Assist Device (LVAD): Any Food and Drug Administration (FDA)-approved LVAD for destination therapy.
Period: Overall Study
Arm/Group | HeartWare® Ventricular Assist System (VAS) | Control Left Ventricular Assist Device (LVAD)
Started | 308 | 157
Completed | 304 | 155
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- HeartWare® VAS: HeartWare® VAS: The HeartWare® VAS is an implantable centrifugal pump that was designed to provide flows up to 10 L/min in a small device that is both lightweight and simple to use.
- Total: Total of all reporting groups
Arm/Group | HeartWare® VAS | Control LVAD | Total
Number analyzed (Participants) | 308 | 157 | 465
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (11.44) | 64.2 (11.14) | 63.6 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 32 | 88
  Male | 252 | 125 | 377
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 3 | 23
  Not Hispanic or Latino | 288 | 154 | 442
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian/Alaska Native | 2 | 1 | 3
  Race: Asian | 1 | 2 | 3
  Race: Black/African American | 72 | 33 | 105
  Race: Native Hawaiian/Pacific Islander | 1 | 0 | 1
  Race: White | 221 | 118 | 339
  Race: Other | 11 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Neurologic Injury
Description: The primary endpoint is the percent of participants at 12 months on the originally implanted device with neurologic injury, defined as a stroke with Modified Rankin Scale (MRS) > 0 at 24-weeks post-stroke, or a transient ischemic attack (TIA), or a spinal cord infarction (SCI). The Modified Rankin Scale is scored from 0 to 6, where 0 indicates an absence of symptoms and 6 indicates death. A score of 4 or higher indicates moderately severe or greater disability.
Time Frame: Implant to 12 Months
Population: Subjects were excluded if they withdrew, were lost to follow-up or have missing outcomes on original device.
Measure: Count of Participants; unit: Participants
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 306 | 157
Participants | 45 | 19
Statistical Analysis 1: Comparison: HeartWare® VAS vs Control LVAD; The primary endpoint is a non-inferiority test comparing HeartWare® VAS to Control; Test type: Non-Inferiority — A non-inferiority margin of 6% was pre-specified; p = 0.1444, Farrington-Manning asymptotic test; Risk Difference (RD) = 2.6, 90% CI 2-sided [-5.5 to 10.7] — Difference = HeartWare® VAS incidence rate - Control incidence rate Two-sided 90% exact binomial confident interval is used

2. Secondary Outcome: Number of HeartWare VAS Participants With Stroke/TIA
Description: The first secondary endpoint is the number of HeartWare VAS participants with stroke/TIA at 12 months on the originally implanted device.
Time Frame: Implant to 12 Months
Population: Subjects were excluded if they withdrew or were lost to follow up on the original device.
Measure: Count of Participants; unit: Participants
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 307
Participants | 59
Statistical Analysis 1: Comparison: HeartWare® VAS; The first secondary endpoint is the percent of participants with stroke/TIA at 12 months on the originally implanted device. It will be compared to 17.7%, which is the lower bound of a pre-defined margin of superiority based on the Endurance clinical trial; Test type: Superiority; p = 0.7363, Exact Binomial Test; Percent of Participants = 19.2, 90% CI 2-sided [15.6 to 23.3] — Two-sided exact binomial confidence interval used

3. Secondary Outcome: Number of Participants With Stroke-Free Success
Description: Success is defined as alive on the originally implanted device, electively transplanted or explanted due to subject recovery and free from disabling stroke (Modified Rankin Scale >=4).
Time Frame: Implant to 12 Months
Population: Subjects were excluded if they had no associated 24 week post-stroke Modified Rankin Scale value, or if the subject withdrew or was lost to follow-up on original device, and no other failure outcome occurred within 1 year post original implant.
Measure: Count of Participants; unit: Participants
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 301 | 157
Participants | 229 | 105
Statistical Analysis 1: Comparison: HeartWare® VAS vs Control LVAD; Test type: Non-Inferiority — The non-inferiority margin on the difference in success proportions is 15%; p < 0.0001, Farrington-Manning asymptotic test; Difference in Percentages = -9.2, 90% CI 2-sided [-17.2 to -1.1] — Difference = Control success rate - HeartWare® VAS success rate Two-sided 90% exact binomial confidence interval is used
Statistical Analysis 2: Comparison: HeartWare® VAS vs Control LVAD; Test type: Superiority; p = 0.0354, Chi-squared

ADVERSE EVENTS:
Time Frame: The adverse events are summarized from the date of implant through 12 months while on the originally implanted device. Subjects are analyzed based on the device they actually received.
Description: The Intermacs (Interagency Registry for Mechanically Assisted Circulatory Support) adverse event definitions are geared towards subjects who have a mechanically circulatory support device.
Groups:
- HeartWare® VAS: Implant of HeartWare® Ventricular Assist System
  HeartWare® VAS: The HeartWare® VAS is an implantable centrifugal pump that was designed to provide flows up to 10 L/min in a small device that is both lightweight and simple to use.
Arm/Group | HeartWare® VAS | Control LVAD
All-Cause Mortality (participants affected / at risk) | 56/308 | 31/157
Serious Adverse Events (participants affected / at risk) | 295/308 | 152/157
Other Adverse Events (participants affected / at risk) | 95/308 | 40/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartWare® VAS (N=308) | Control LVAD (N=157)
Major Bleeding (Blood and lymphatic system disorders) | 156 (297) | 87 (190)
Cardiac Arrhythmia (Cardiac disorders) | 95 (132) | 42 (49)
Device Malfunction/Failure (Product Issues) | 60 (81) | 38 (46)
Hemolysis (Blood and lymphatic system disorders) | 3 (4) | 8 (8)
Hepatic Dysfunction (Hepatobiliary disorders) | 10 (10) | 6 (6)
Hypertension (Cardiac disorders) | 27 (34) | 12 (12)
Major Infection (Infections and infestations) | 150 (259) | 85 (149)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2)
Neurological Dysfunction (Nervous system disorders) | 57 (83) | 24 (26)
Pericardial Fluid Collection (Cardiac disorders) | 17 (18) | 13 (15)
Psychiatric Episode (Psychiatric disorders) | 34 (35) | 11 (12)
Renal Dysfunction (Renal and urinary disorders) | 32 (35) | 23 (25)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 61 (74) | 31 (37)
Right Heart Failure (Cardiac disorders) | 94 (101) | 56 (61)
Arterial Non-CNS Thromboembolism (Vascular disorders) | 3 (3) | 0 (0)
Venous Thromboembolism (Vascular disorders) | 11 (11) | 4 (5)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Other Intermacs (General disorders) | 219 (599) | 106 (265)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartWare® VAS (N=308) | Control LVAD (N=157)
Cardiac Arrhythmia (Cardiac disorders) | 16 (19) | 7 (7)
Device Malfunction/Failure (Product Issues) | 18 (26) | 1 (1)
Hypertension (Cardiac disorders) | 16 (20) | 8 (9)
Major Infection (Infections and infestations) | 33 (41) | 24 (32)
Other Intermacs (General disorders) | 29 (30) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, the contract allows the principal investigator to publish their data after the release of the multi-center publication (or one year after the conclusion of the study if no multi-center publication is submitted) following the sponsor review for (a) disclosure of confidential information, and (b) information that would impair the sponsor's ability to obtain patent protection.